CLINICAL TRIAL: NCT07204730
Title: Comparing the Effect of Peer Group Training and Direct Instruction on Mechanisms to Counteract Cyberbullying Among Male High School Students in Tehran
Brief Title: Peer Group Training vs Direct Instruction to Reduce Cyberbullying Among High School Boys"
Acronym: CyberPeer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fereshteh Javanmardi, PhD, Principal Investigator, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ORG-2025-001; CB-TEHRAN-2025 (Other: Dept. Social Medicine, Ahvaz Jundishapur Univ. Med. Sci.)
Record Dates: First submitted 2025-09-13; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cyberbullying
Keywords: Cyberbullying; Peer Education; Social Skills Training; Emotional Intelligence; High School Students; Adolescent Behavior; Virtual Harassment; School-based Intervention; Peer-led Training; Direct Instruction
MeSH Terms: conditions — Cyberbullying; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three groups: direct psychologist-led training, peer-mediated training, or control (no intervention). Each group received its assigned intervention (or no intervention) simultaneously, and outcomes were assessed at baseline and three months post-intervention to compare effectiveness across groups.
Masking Description: This study was conducted as an open-label trial. Neither the participants, the peer or psychologist trainers, nor the outcome assessors were blinded to group assignments. All parties were aware of which intervention each participant received, as blinding was not feasible for this behavioral and educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct Psychologist-Led Training (Experimental): participants received six two-hour social skills training sessions delivered directly by a licensed psychologist. The sessions focused on problem-solving, empathy, stress management, and strategies to counteract cyberbullying. Outcomes were assessed at baseline and three months post-intervention.
  Interventions: Behavioral: Direct Social Skills Training
- Peer-Mediated Training (Experimental): A small volunteer group of students attended six two-hour sessions with a psychologist and then delivered the same curriculum to their peers. Weekly progress reports were submitted to the psychologist to ensure fidelity. Emotional intelligence and cyberbullying outcomes were measured at baseline and three months post-intervention.
  Interventions: Behavioral: Peer-Led Social Skills Training
- Control Group (Sham Comparator): Participants received no training during the study period. Outcomes were measured at baseline and three months post-intervention to serve as a comparison for the intervention groups.
  Interventions: Other: Control No Training

INTERVENTIONS:
Behavioral: Direct Social Skills Training — Participants attended six two-hour sessions led by a licensed psychologist. Sessions focused on social skills, including empathy, problem-solving, stress management, and strategies to prevent and counteract cyberbullying. Outcomes were measured at baseline and three months post-intervention.
  Arms: Direct Psychologist-Led Training
Behavioral: Peer-Led Social Skills Training — A volunteer group of students attended six two-hour sessions with a psychologist and then taught their peers the same curriculum. Weekly progress reports were submitted to the psychologist to ensure fidelity. Outcomes on emotional intelligence and cyberbullying were assessed at baseline and three months post-intervention.
  Arms: Peer-Mediated Training
Other: Control No Training — Participants in the control group received no intervention during the study period. Outcomes were assessed at baseline and three months post-intervention to provide a comparison for the experimental groups.
  Arms: Control Group

SUMMARY:
This study aims to explore ways to reduce cyberbullying among male high school students in Tehran by comparing two types of training: direct instruction from a psychologist and peer-led training. Cyberbullying is a serious problem that affects many teenagers, causing stress, emotional difficulties, and social challenges. Learning effective strategies to prevent and respond to cyberbullying may help improve students' emotional skills and overall well-being.

The study includes 252 male students from grades 9 to 11 in three high schools. School staff first attend a short session to learn about cyberbullying and its consequences. Students are then randomly assigned to one of three groups:

Direct Training Group: A psychologist leads six two-hour sessions teaching social skills such as empathy, problem-solving, and stress management.

Peer Training Group: A smaller group of volunteer students attends the same sessions and then shares the information with their classmates. Their progress is monitored weekly.

Control Group: Students receive no special training.

Assessments are conducted before the program and three months after it ends. All students complete a questionnaire that measures emotional intelligence and experiences with cyberbullying.

This study will provide information on the design, implementation, and feasibility of social skills training programs aimed at addressing cyberbullying in high school settings.

DETAILED DESCRIPTION:
The rapid growth of Internet use among adolescents has introduced both opportunities and risks. One significant concern is cyberbullying, defined as intentional, repeated harm inflicted through electronic communication. Male high school students may be particularly vulnerable to engaging in or being targeted by cyberbullying, and schools often lack structured programs to address these behaviors. Previous research suggests that social skills training, including empathy development, problem-solving, and stress management, may improve emotional regulation. Peer-led interventions have also been proposed as a strategy to leverage social influence to reinforce positive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Male students in grades 9-11.

Age between 15 and 20 years.

Enrolled in one of the participating high schools in Tehran.

Parental/guardian consent and student assent provided.

Willingness to participate in training sessions and complete questionnaires.

Exclusion Criteria:

* Prior participation in intensive social skills or anti-cyberbullying training programs.

Diagnosed psychological disorders that would interfere with participation.

Inability to attend intervention sessions or follow-up assessments.

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 252 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Emotional Intelligence | Baseline (pre-test) and theree months post-intervention
  Emotional intelligence will be measured using the Bar-On Emotional Intelligence

SECONDARY OUTCOMES:
Cyberbullying Roles (Bully, Victim, Both, Neither) | Baseline (pre-test) and three months post-intervention
  Emotional intelligence will be assessed using the Bar-On Emotional Intelligence Inventory (EQ-i), which evaluates intrapersonal, interpersonal, stress management, adaptability, and general mood domains. Scores range from 0 to 100, with higher scores indicating greater emotional intelligence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahvaz Jundishapur University of Medical Sciences, Ahvāz, Iran

IPD SHARING:
Plan to Share IPD: Undecided
At this time, a plan for sharing individual participant data (IPD) has not been finalized. The study involves data from high school students, including sensitive behavioral and emotional information. Any future sharing of data would follow strict de-identification procedures and comply with ethical guidelines and school policies to protect participant privacy.

REFERENCES:
- [Result] Palladino BE, Nocentini A, Menesini E. Evidence-based intervention against bullying and cyberbullying: Evaluation of the NoTrap! program in two independent trials. Aggress Behav. 2016 Mar-Apr;42(2):194-206. doi: 10.1002/ab.21636. PMID 26879897
- [Result] Fousiani K, Dimitropoulou P, Michaelides MP, Van Petegem S. Perceived Parenting and Adolescent Cyber-Bullying: Examining the Intervening Role of Autonomy and Relatedness Need Satisfaction, Empathic Concern and Recognition of Humanness. J Child Fam Stud. 2016;25:2120-2129. doi: 10.1007/s10826-016-0401-1. Epub 2016 Mar 9. PMID 27375346
- [Result] Clonan-Roy K, Jacobs CE, Nakkula MJ. Towards a model of positive youth development specific to girls of color: Perspectives on development, resilience, and empowerment. Gender Issues. 2016; 33:96-121.
- [Result] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Result] Zhu C, Huang S, Evans R, Zhang W. Cyberbullying Among Adolescents and Children: A Comprehensive Review of the Global Situation, Risk Factors, and Preventive Measures. Front Public Health. 2021 Mar 11;9:634909. doi: 10.3389/fpubh.2021.634909. eCollection 2021. PMID 33791270

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT07204730/Prot_SAP_000.pdf